CLINICAL TRIAL: NCT02311634
Title: A Comparison of Efficacies of Electrical Pudendal Nerve Stimulation Versus Transvaginal Electrical Stimulation in Treating Urge Incontinence
Brief Title: A Comparison of Electrical Pudendal Nerve Stimulation and Transvaginal Electrical Stimulation for Urge Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12401904600
Record Dates: First submitted 2014-11-19; First posted 2014-12-08 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2015-06

CONDITIONS: Urge Urinary Incontinence
Keywords: Electrical pudendal nerve stimulation; Transvaginal electrical stimulation; Urge urinary incontinence; Comparative study
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical pudendal nerve stimulation (Experimental): At a frequency of 2.0 Hz and a moderate intensity (25~35 mA); 60 minutes three times a week for a total of three weeks
  Interventions: Device: Electrical pudendal nerve stimulation
- Transvaginal ES (Active Comparator): At a current intensity of < 60 mA (in 5% increments from 0 mA to the intensity that is sensed without obvious discomfort) and frequencies of 12.5 to 30 Hz, 45 min three times a week for a total of four weeks.
  Interventions: Device: Transvaginal ES

INTERVENTIONS:
Device: Electrical pudendal nerve stimulation — Four sacral points are selected. The two upper points are located about 1 cm bilateral to the sacrococcygeal joint. On the upper points, a needle of 0.40 Х 100 mm is inserted perpendicularly to a depth of 80 to 90 mm to produce a sensation referred to the urethra or the anus. The locations of the two lower points are about 1 cm bilateral to the tip of the coccyx. On the lower points, a needle of 0.40 Х 100 or 125 mm is inserted obliquely towards the ischiorectal fossa to a depth of 90 to 110 mm to produce a sensation referred to the urethra. After the sensation referred to the above regions is produced, each of two pairs of electrodes from a G6805-2 Multi-Purpose Health Device is connected with the two ipsilaterally inserted needles.
  Arms: Electrical pudendal nerve stimulation
Device: Transvaginal ES — A neuromuscular stimulation therapy system (PHENIX USB 4，Electronic Concept Lignon Innovation, France) is used for TES
  Arms: Transvaginal ES

SUMMARY:
The purpose of this study is to determine whether electrical pudendal nerve stimulation is more effective than transvaginal electrical stimulation in treating urge urinary incontinence (UUI).

DETAILED DESCRIPTION:
Electrical neuromodulation can be used to treat UUI refractory to medication. Electrical neuromodulation therapies include transvaginal or transanal electrical stimulation (TES), percutaneous tibial nerve stimulation (PTNS), sacral neuromodulation (SNM), and pudendal neuromodulation (PNM). TES is easily applicable but is sometimes intolerable for many patients due to discomfort, mucosal injury, and high-intensity stimulation necessary to obtain acceptable outcome. SNM with the InterStim device differs from TES by its continuous stimulation and close nerve contact. It has a high rate of success, but symptoms appear to recur almost immediately after discontinuation of the stimulation, and at least 20 % of patients initially tested do not respond to a test procedure. Its disadvantages included invasiveness, high cost of treatment, high surgical revision rate, device replacement required when battery runs out, and adverse events. PNM with the Interstim device or the Bion device can be used to treat UUI refractory to SNM, but this therapy also has the disadvantages similar to those of SNM. PTNS with needle electrodes is minimally invasive, demonstrates efficacy, and is easily applicable and well tolerated, but PTNS effects diminish over time after the end of treatment.

By combining the advantages of PTNS and PNM and incorporating the technique of deep insertion of long acupuncture needles, the investigators developed electrical pudendal nerve stimulation (EPNS). In EPNS, long acupuncture needles of 0.40 Х 100 or 125 mm were deeply inserted into four sacral points and electrified to stimulate the pudendal nerves (PN). CT transverse plane at the coccygeal apex has showed that the position of the lower needle tip is similar to where (adjacent to PN at Alcock's canal) the Bion device is implanted for chronic PN stimulation. Besides the radiographic evidence, simultaneous records of perineal ultrasonographic pelvic floor muscle contraction, vaginal pressure and pelvic floor surface electromyogram in our previous study have proved that EPNS can exactly excite PN. The purpose of this study is to compare the efficacies of EPNS versus TES in treating female UUI.

ELIGIBILITY:
Inclusion Criteria:

* UUI history
* Positive pad test result
* Urodynamic study: A decrease in bladder capacity at the first desire for urination; a decrease in maximum bladder capacity; low compliance bladder

Exclusion Criteria:

* UUI that can be relieved by drugs
* Neurogenic or non-neurogenic UUI
* Other types of incontinence such as stress incontinence and overflow incontinence

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
A questionnaire to measure the severity of UUI symptoms | three or four weeks
24-hour urine leakage amount | three or four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Siyou Wang, Master, Study Chair — Shanghai research institute of acupuncture and meridian
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China

REFERENCES:
- [Result] Wang S, Zhang S, Zhao L. Long-term efficacy of electrical pudendal nerve stimulation for urgency-frequency syndrome in women. Int Urogynecol J. 2014 Mar;25(3):397-402. doi: 10.1007/s00192-013-2223-7. Epub 2013 Oct 3. PMID 24091564